CLINICAL TRIAL: NCT00508807
Title: Clinical Study Protocol RTA 402-C-0501: A Phase I Dose-finding and Pharmacokinetic Study of RTA 402 (CDDO-Me) Administered Orally for 21 Days of a 28-day Cycle in Patients With Advanced Solid Tumors or Lymphoid Malignancies
Brief Title: RTA 402 in Advanced Solid Tumors or Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Reata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0984
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoid Malignancies; Solid Tumors
Keywords: Lymphoid Malignancies; Solid Tumors; RTA 402

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RTA 402 (Experimental): 5 mg PO daily x 21 days
  Interventions: Drug: RTA 402

INTERVENTIONS:
Drug: RTA 402 — 5 mg by mouth (PO) daily for 21 days

SUMMARY:
Primary:

* To determine the dose-limiting toxicity, maximum tolerated dose, and recommended phase II dose of RTA 402 capsules in patients with advanced solid tumors or lymphoid malignancies who have failed standard-of-care curative or survival-prolonging therapy, or for whom no such therapies exist.
* To characterize the pharmacokinetics of RTA 402 capsules administered orally for 21 days in this patient population.

Secondary:

* To document any preliminary antitumor activity of RTA 402 in this patient population.
* To determine the in vivo molecular and biological effects of RTA 402 by measuring changes in markers of differentiation, apoptosis, and anti-inflammatory effects in WBCs, blood plasma, and, in consenting patients, tumor biopsies.
* To correlate the biological activity of RTA 402 with drug concentration in plasma and blood cellular elements
* To evaluate the series of inflammation related symptoms over the course of the study, and to determine the correlation of symptom intensity with plasma cytokines.

DETAILED DESCRIPTION:
RTA 402 is a new man-made drug that is designed to inhibit (turn off) genes that may activate your cancer cells and cause them to grow. This drug has not been tested in humans.

If you are found to be eligible to take part in this study, you will take RTA 402 by mouth (several capsules a day) in the morning with a glass of water (before eating) on the dose level that will be assigned to you. The dose level you receive will depend on when you begin on this study. You will receive the study drug for 21 days in a row. You will not take the study drug for the next 7 days. This is considered a rest period. These 28 days equal 1 cycle. You should take your study drug as instructed. If a dose is missed or vomited, it will not be replaced either on that day or at the end of the 21-day treatment period.

At the beginning of the study, one to three patients may be enrolled at each dose level, and dose will be doubled between groups until the first occurrence of intolerable side effects during Cycle 1. At the first occurrence of less severe side effects, groups will be expanded to 3-4 patients. Dose escalation (increasing) will continue in this way until researchers learn the highest dose that is best tolerated. You will remain at the same dose level that you started on for at least 2 cycles. After at least 2 cycles, your dose may be increased to another dose that has been determined to be safe. If your disease gets worse or you experience any intolerable side effects, you will be taken off this study.

On Cycle 1 on Days 1 and 21, you will be asked to go to the Clinical and Translational Research Center for your dose of the study drug. You will be asked about how you are feeling, and about any medications you may be taking including any over the counter medication, herbs, and alcohol. You will be asked to report any bad side effects you may experience from the study drug. You will have blood draws (about 1 1/2 teaspoons each time) for PK studies. You will have these PK blood draws before you take RTA 402 at 15 minutes, 30 minutes, and 1, 2, 4, 6, 8, and 24 hours after you take the study drug. You will have your vital signs measured at 2, 4, and 8 hours after taking RTA 402. You will have your urine collected over a 24-hour period. The study staff will provide the urine sample container and explain how to collect your urine.

During Cycle 1, you will return to the clinic every week to have routine blood drawn (about 2 teaspoons) to check the status of your disease. You will be asked how you are feeling and about any medications you may be taking including any over the counter medication, herbs, and alcohol.

Each week during Cycle 1 and on Day 28 of each additional cycle, you will complete 2 questionnaires that will take about 15 minutes to complete. You will also have your body weight measured and be asked about your normal food intake. Your body composition will be measured using measurements that include body weight and height, skin fold thickness, and bioelectrical impedance using the Tanita body composition monitoring scale. This is a non-invasive method to measure total body water, total body fat, and total body lean mass. Researchers will measure how much energy your body uses while at rest. You will also have timed test that will involve your participation where at your fastest speed you will be asked to walk 25 feet and walk back.

After Cycle 1, you will return to the clinic every other week for up to 18 cycles (about 18 months) as long as your health does not get worse and you do not experience any intolerable side effects.

During every other cycle starting with Cycle 2, you will be evaluated to check the status of your cancer. You will have routine imaging studies, such as x-rays, CT scans, or MRIs to measure your tumor. You will have a bone marrow biopsy (if you have lymphoid disease) to measure your disease. On Day 1 of the next cycle, you will return to your doctor's office for your next physical exam and to begin the next cycle of the study drug.

While on this study, you will not be allowed to take any other investigational agent, chemotherapy, biologic therapy, immunotherapy, or anti-cancer treatments. You will not be allowed to take medicine that can help increase your white blood cell count.

Once you have completed all cycles of the study drug, you will have an end-of-study visit. During this visit, you will have a physical exam, including measurement of your vital signs. You will have blood drawn (about 1 1/2 teaspoons) for routine tests, and a urine sample will be collected. You will have a bone marrow biopsy (if you have lymphoid disease) to measure your disease. You will have imaging studies, such as x-rays, CT scans, or MRIs to measure your tumor. You will be asked to report any side effects or new medications that you may be taking including any over the counter medication, herbs, and alcohol.

You will be followed (30 days after you are off study) and asked to report any side effects you may be experiencing, or new medications that you may be taking. You will also have a physical exam, including measurement of your vital signs. If your doctor thinks that you should continue taking RTA 402 (after 18 cycles or 18 months), you will be asked to participate in an extended study.

This is an investigational study. RTA 402 has been authorized by the FDA for use in research only. Up to 45 patients will take part in this multicenter study. Up to 42 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion:

1. Age >/= 18 years
2. Patient must have histopathological documentation of solid tumor or lymphoid malignancy. (measurable disease is not required)
3. Patient must have advanced or metastatic cancer that are either refractory or has relapsed after standard-of-care curative or survival-prolonging therapy, or for whom no such therapies exist. (there is no limit on the number of prior lines of therapy)
4. Patient must be ECOG performance status of less than or equal to 2.
5. Patient must have adequate liver and renal function as documented by the following laboratory test results within 14 days of starting therapy:

   * total bilirubin </= 1.5 mg/dL
   * AST (SGOT) and ALT(SGPT) </= 2.5 ULN or
   * </= 5 ULN if liver is involved by tumor
   * creatinine </= 2.0 mg/dL OR creatinine clearance > 60 mL/min
6. Patient must have adequate bone marrow function as documented by the following laboratory test results within 14 days of starting therapy:

   * platelets greater than 100,000/mm^3,
   * absolute granulocyte count greater than 1,500/mm^3,
   * hemoglobin greater than or equal to 8.0 g/dl.
7. Patient must have completed prior chemotherapy, hormonal therapy, radiation therapy, biological therapy, or other investigational cancer therapy at least 4 weeks prior to starting RTA 402, and must have recovered from all acute side effects (to CTC grade 1 or less) prior to initiation of RTA 402. Patients who were receiving mitomycin C or nitrosoureas must be 6 weeks from the last administration of chemotherapy.
8. Patient (man or woman) must agree to practice effective contraception during the entire study period unless documentation of infertility exists.
9. Patient must have a life expectancy of more than 3 months.
10. Patient must be able and willing to sign the informed consent form.
11. Patient must be willing and able to self-administer orally and document all doses of RTA 402 ingested.

Exclusion:

1. Patients with active brain metastases or primary CNS malignancies. (patients with a previously treated brain metastasis may be included)
2. Patients who are pregnant or breast feeding
3. Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to:

   * uncontrolled diabetes
   * active or uncontrolled infection
   * acute or chronic liver disease (i.e., hepatitis, cirrhosis)
   * confirmed diagnosis of HIV infection
   * uncontrolled hypertension, symptomatic congestive heart failure,
   * unstable angina pectoris,
   * myocardial infarction within the past 6 months, or
   * uncontrolled cardiac arrhythmia.
4. Patients with psychiatric illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of RTA 402 | 28 day cycles

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org